CLINICAL TRIAL: NCT07009522
Title: Hamburg Emotion Awareness and Regulation Group Training for Autistic Adolescents (HEART)
Acronym: HEART
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johannes Boettcher, Research group leader and principle investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPEK-0914; 04/107 (Other Grant/Funding Number: Werner Otto Stiftung)
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Study Group

STUDY DESIGN:
Intervention Model Description: The study design is group-based intervention with a one-arm design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): study group
  Interventions: Behavioral: Hamburg Emotion Awareness and Regulation Group Training for Autistic Adolescents - HEART

INTERVENTIONS:
Behavioral: Hamburg Emotion Awareness and Regulation Group Training for Autistic Adolescents - HEART — The group program for adolescents with ASD takes place weekly. Each session lasts 100 minutes (including a break), and the training includes a total of 12 sessions. The intervention is manualized and is based on the theoretical foundations of Cognitive Behavioral Therapy, Mindfulness-Based Therapy, and the TEACCH approach (Mesibov et al., 2005). Parallel to the adolescents, their parents will participate in a separate group training, which will be conducted in five sessions of 100 minutes each and is closely linked in content to the adolescent group training.

SUMMARY:
The study focuses on a group training program called HEART aimed at helping adolescents with Autism Spectrum Disorder improve emotional regulation. It will use a pilot trial to evaluate the program's feasibility and effectiveness. The findings aim to advance scientific understanding and support the development of effective, evidence-based interventions to strengthen psychosocial support for autistic adolescents.

DETAILED DESCRIPTION:
Adolescents with Autism Spectrum Disorder (ASD) often experience significant difficulties in emotional regulation due to increasing developmental challenges, which can lead to a higher prevalence of psychological comorbidities such as anxiety disorders and depression. Despite the urgent need for specific therapeutic interventions, this area remains largely underrepresented in clinical practice and research. The present study aims to address this gap by investigating the feasibility and effectiveness of the behavioral therapy program "Hamburg Emotion Awareness and Regulation Group Training for Autistic Adolescents (HEART). A pilot trial will be used to evaluate the feasibility and acceptability of the intervention. The intervention group will participate in a group training adapted to the needs of adolescents with ASD. This pilot study could significantly contribute to the scientific understanding of emotion regulation in adolescents with ASD and support the development of practically relevant evidence-based interventions. The study's findings could have important implications for clinical practice. The group training is based on proven behavioral therapy methods established among therapists in Germany. The manualized manual for the adapted application of these methods with autistic adolescents could thus serve as a foundation for improving psychosocial care for this target group.

ELIGIBILITY:
Autistic adolescents will be included in the study, recruited from various departments of the Clinic for Child and Adolescent Psychiatry, Psychotherapy, and Psychosomatics at UKE, as well as from autism therapy centers. Eligible participants are adolescents aged 13 to 18 years who meet the criteria for a primary diagnosis of an autism spectrum disorder-including early childhood autism (ICD-10: F84.0), atypical autism (ICD-10: F84.1), and Asperger's syndrome (ICD-10: F84.5)-and who have sufficient knowledge of the German language. The diagnosis should be confirmed based on developmental history, the ADOS-2 assessment, and a clinical diagnosis from a specialized clinician. Additionally, only autistic adolescents exhibiting difficulties in emotion regulation (measured by the Emotion Regulation Inventory (EDI-SF), T-score ≥ 60) will be included. Exclusion criteria are: below-average cognitive abilities, IQ ≤ 85 (ICD-10: F70); lack of German language skills; or significant visual or hearing impairments that cannot be corrected. Furthermore, patients with severe neurological or psychiatric conditions (e.g., epilepsy, syndromic disorders with neuropsychiatric involvement, psychoses) or current acute suicidality, as assessed clinically, will be excluded.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Emotion Dysregulation | Lead-in period" (6 weeks before randomization; T0); start ("Baseline," T1) and end (T2) of the treatment, as well as 6 weeks (T3) and 12 weeks (T4) after the completion of the 3-month intervention.
  The Emotion Dysregulation Inventory - Short Form (EDI-SF, Mazefsky, Day, et al., 2018; Mazefsky, Yu, et al., 2018) is a 13-item questionnaire designed to assess emotion regulation problems in children and adolescents through self-report and parent-report. The items are answered on a five-point Likert scale, ranging from 1 = "not at all" to 5 = "very severe." The questionnaire evaluates two scales: "Reactivity" and "Dysphoria." Higher scores indicate greater emotional dysregulation. The primary outcome criterion is emotion regulation, which will be assessed from the parent perspective using the EDI-SF.

SECONDARY OUTCOMES:
Autistic Traits | Lead-in period" (6 weeks before randomization; T0)
  The Social Responsiveness Scale (SRS-16; Constantino et al., 2003) is a quantitative measure of autistic traits in children, adolescents, and adults. The SRS-16 (Sturm et al., 2017) is a 16-item parent questionnaire designed to assess social, communicative, and rigid behaviors in children and adolescents for dimensional autism diagnostics. The items are answered on a four-point response scale, ranging from 1 = "not at all" to 4 = "almost always." A total score is calculated by summing the items. The total score ranges from 16 to 80, with higher values indicating greater severity of impairment. The SRS has demonstrated good psychometric properties and cross-cultural validity for the assessment of ASD (Bölte et al., 2008, 2011).
Quality of Life and psychological well-being | Lead-in period" (6 weeks before randomization; T0); start ("Baseline," T1) and end (T2) of the treatment, as well as 6 weeks (T3) and 12 weeks (T4) after the completion of the 3-month intervention
  The KIDSCREEN-10 (Ravens-Sieberer et al., 2010) is a brief, standardized instrument for assessing the quality of life and psychological well-being of children and adolescents aged 8 to 18 years from self-report and parent perspective. The KIDSCREEN-10 includes a total of 10 items focusing on various dimensions of quality of life, including emotional well-being, social well-being, physical health, and joy of life. The items are answered on a five-point response scale, ranging from 1 = "not at all true" to 5 = "completely true." The questionnaire is characterized by good psychometric validity and reliability and is suitable for use across different populations (Ravens-Sieberer et al., 2010).
Self-perceived depressive symptoms | Lead-in period" (6 weeks before randomization; T0); start ("Baseline," T1) and end (T2) of the treatment, as well as 6 weeks (T3) and 12 weeks (T4) after the completion of the 3-month intervention
  The Beck Depression Inventory for Youth - Second Edition (BDI-Y-2; Beck et al., 2001) is a self-report questionnaire designed to assess the severity of depressive disorder in children and adolescents aged 7 to 18 years. For adults aged 18 and above, the Beck Depression Inventory-II (BDI-II) is used. The 20 items measure negative thoughts of the child or adolescent about themselves, their life, and the future, as well as feelings of sadness and physiological symptoms of depression, based on the diagnostic criteria of DSM-5. The German version of the instrument demonstrates acceptable psychometric properties (Beck et al., 2001; Siefen & Busch, 2018).
Self-perceived anxiety symptoms | Lead-in period" (6 weeks before randomization; T0); start ("Baseline," T1) and end (T2) of the treatment, as well as 6 weeks (T3) and 12 weeks (T4) after the completion of the 3-month intervention
  The Beck Anxiety Inventory for Youth - Second Edition (BAI-Y-2; Beck et al., 2001) is a self-report questionnaire designed to assess the severity of anxiety in children and adolescents aged 7 to 18 years. For adults aged 18 and above, the Beck Anxiety Inventory (BAI) is used. The 20 items assess specific and generalized anxieties, including fears related to school, fear of injury, and health-related anxieties. Additionally, the inventory captures various symptoms of anxiety, such as rumination and worry-driven thoughts, as well as physiological symptoms, based on the diagnostic criteria of DSM-5. The German version of the instrument demonstrates acceptable psychometric properties (Beck et al., 2001; Siefen & Busch, 2018).
Quality of Parent-Adolescent Communication | Lead-in period" (6 weeks before randomization; T0); start ("Baseline," T1) and end (T2) of the treatment, as well as 6 weeks (T3) and 12 weeks (T4) after the completion of the 3-month intervention
  The Parent-Adolescent Communication Scale (PACS; Barnes & Olson, 1982) is a questionnaire used to assess the quality of dyadic parent-child communication between parents and adolescents. The PACS is available for self-report and third-party assessment and includes the subscales "Open Communication" and "Communication Problems." The short version of the instrument contains 6 items, which are answered on a five-point response scale from 1 = "strongly disagree" to 5 = "strongly agree." The problematic items are recoded afterward. The sum of the items is calculated to obtain a total score, which ranges from 6 to 30, with higher scores indicating better quality of parent-child communication. The German version of the PACS demonstrates good psychometric properties (Zapf & Boettcher, 2024).
Patient satisfaction | (T4) after the completion of the 3-month intervention
  The Questionnaire for Patient Satisfaction (ZUF-8; Schmidt et al., 1989) is an instrument used to assess overall patient satisfaction at the end of an intervention. The ZUF-8 comprises eight items, which are answered on a four-point Likert scale. The total score is calculated by summing the items, resulting in a score ranging from 8 to 32, with higher values indicating greater patient satisfaction. There are both an adult version for parents and a child version. The ZUF-8 demonstrates good psychometric properties (Kriz et al., 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Boettcher, Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf

IPD SHARING:
Plan to Share IPD: No